CLINICAL TRIAL: NCT03638622
Title: Low-cost Enabling Technology for Image-guided Photodynamic Therapy (PDT) of Oral
Brief Title: Low-cost Enabling Technology for Image-guided Photodynamic Therapy (PDT) of Oral Cancer Cancer.
Acronym: UH3-India
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Jawaharlal Nehru Medical College (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tayyaba Hasan,Ph.D., Professor of Dermatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001855; 5UH3CA189901-04 (NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Oral Cancer
Keywords: Oral cancer, Photodynamic Therapy, Photosensitizer, ALA
MeSH Terms: conditions — Mouth Neoplasms | interventions — Photochemotherapy; Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Trial with single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aminolevulinic acid (ALA) and Photodynamic Therapy (PDT) (Experimental): Aminolevulinic Acid (ALA) administration, Photodynamic Therapy (PDT) treatment using LED (Light-emitting diode) light source and follow-up.
  Interventions: Combination Product: Photodynamic Therapy

INTERVENTIONS:
Combination Product: Photodynamic Therapy — Patients receive aminolevulinic acid (ALA) orally with orange juice in 3 fractions at 0,1,2 hours before undergoing photodynamic therapy using LED based Device on day one.
  Other Names: Aminolevulinic acid (ALA); Photodynamic Therapy (PDT); Light Emitting Diode (LED) based Device

SUMMARY:
Oral cancer in India affects mostly those from the lower socioeconomic groups, due to a higher exposure to risk factors such as the use of tobacco, zarda, khaini, chewing gutka, mawa, and kharra, which are all dry mixtures of flavorings, areca nut flakes and powdered tobacco. Earlier detection of oral cancer offers the best chance for long-term survival and has the potential to improve treatment outcomes and make healthcare affordable. Current treatment options, primarily surgery and/or radiation, can be curative if cancer or dysplasia is caught at a sufficiently early stage. Though even in these cases treatment may be disfiguring with significant impact upon quality of life, and many patients do not seek medical attention until the disease has progressed to a point where radical operation is required (Stage III/IV), often entailing block dissection and removal of the entire lymphatic drainage of the neck. Despite the radical operation, the disease still recurs, leading to an overall survival rate of less than 70% of these cases. The present study evaluates photodynamic therapy (PDT) as an alternative intervention for early-stage malignant lesions of the oral cavity using a low-cost and battery-powered platform that is specifically adapted for low and middle-income countries (LMIC) implementation.

DETAILED DESCRIPTION:
Study Facility:

Pre-study Screening: Patients come to Ear, Nose, and Throat (ENT)/Oral and Maxillofacial/Plastic and Reconstructive surgery outpatient facilities. Typically, an ENT specialist handles early cases (biopsy proven malignancies), while ENT and plastic surgeons jointly deal with advanced cases. Patients screening will take place in outpatient departments. The investigator/s will interview each subject to develop a brief, relevant medical history and determine that all selection criteria are met. The subject will receive an explanation of the study objectives, possible risks and benefits of the study. After history evaluation of the patients, Blood work will be done to check liver functions Test. After the blood report and inclusion and exclusion criteria, the consultant will discuss and educate the patients about photosensitization and Photodynamic Therapy (PDT). If patients are willing to take part in the study, co-investigator will obtain a signed consent form. After obtaining a signed consent form, the consultant will schedule an appointment for PDT therapy.

Procedure after enrollment: Investigators plan to enroll 30 patients with oral cancer in this study. The study will take place at Jawaharlal Nehru Medical College (JNMC), Aligarh. This timeline of procedures considers that many patients may need to travel from remote rural areas with poor access to transportation, so it cannot be assumed that patients have convenient access to return to the clinic for multiple repeated biopsies.

Aminolevulinic Acid (ALA) preparation and administration: The FDA-approved Aminolevulinic Acid (ALA) from Dusa Pharmaceuticals, Inc., Wilmington, Massachusetts (MA) will be used in powder form. Patients will initially receive a baseline ultrasound of the oral cavity prior to ALA administration. In the case of potentially childbearing women, a serum pregnancy test will be performed before ALA administration by SD (Standard Diagnostic Inc, India) Bioline kit. One hour prior to ALA administration, analgesic (Aceclofenac 200mg, Intas Pharmaceuticals, India), anti-inflammatory drug (HifenacSR 200mg; Intas Pharmaceuticals, India) and antiemetic (Domperidone, Domperon, 10mg; Cadila Pharmaceuticals, Inc., India) will be given to patients orally to avoid nausea and pain. ALA, totaling 60 mg/kg, will be administered orally via three repeated doses of 20 mg/kg of ALA dissolved in either orange juice or a soft drink, which lowers the potential of hydrogen (pH) of the solution, at 0, 1 and 2 hours.

Day One: Baseline imaging; Fluorescence measurement: PpIX (Protoporphyrin IX) fluorescence will be recorded using 405nm excitation light delivered from an Light-Emitting Diode (LED) source powered by a smartphone. This is a non-invasive system. The PpIX fluorescence will be photographed using the camera embedded in the smartphone. The advantage of this step is that in the long term it will obviate the need for biopsies to establish PpIX concentrations and could allow for online dosimetry customized to individual patients. Three photographs will be taken in each subject: first photograph will be taken prior to given ALA to the patients, second photograph after 2-3 hours of ALA incubation, and third photograph will be taken immediately after PDT treatment.

Imaging Procedure before treatment: After allowing 2-3 hours for PpIX conversion and accumulation in the malignant tissue, a baseline image of the tumor will be obtained using the smartphone PpIX imaging approach. In this clinical validation study, these PpIX fluorescence images will be used to make treatment decisions beyond visual guidance for applicator placement on the lesion.

PDT Procedure: Immediately after the brief imaging session (approximately 5 minutes), the PDT treatment will proceed. Depending on the exact fractionation schedule determined, a total fluence of 100Joule/cm2 at the lesion surface will be delivered with an area of applicators or compressed applicator in for approximately 30-45 minutes. Placement will be such that the full extent of the lesion falls within a 1mm margin of the applicator area. Every 10 minutes, a 2-3 minute break is provided to the patient and the study personal will check for the correct placement of the probe. The clinician will conduct applicator placement with the assistance of a nurse as needed so that it fits tightly in contact with the active surface facing the lesion. Care will be required when pressing an applicator tipped light delivery system hard against tissue. If one press too hard and the tissue is rendered temporarily hypoxic, there will be no PDT effect. During therapy patients will leave their mouth closed around the optical fiber. Depending on the exact orientation of the lesion within the oral cavity a mouth guard may be used to aid applicator positioning, or if this improves patient comfort. Also, to aid in the stabilization of the fiber and improve patient comfort, an ergonomic external positioning mount may be employed to help maintain the optical fiber in position. Provided that care is taken that no incidental body movements during irradiation lead to significant shifting of movement of the applicator, patients will be able to read a magazine, watch television (TV) if available or other similar activities from a seated position. Small lesions may receive a complete treatment in this time interval, while (as noted above), larger lesions may require one or more additional applications. Patients will receive analgesic Aceclofenac, HifinacSR (200 mg); Intas Pharmaceuticals, India to avoid pain. Appropriate Laser safety glasses will also be provided to the patients during irradiation.

Post-treatment imaging: At the conclusion of the PDT treatment, the light delivery fiber will be removed and a follow-up smartphone fluorescence image will be obtained for later analysis of PpIX photobleaching. Patients will receive guidance on the resumption of normal activities. After the procedure, patient will be advised to avoid foods that are spicy, hot or oily for at least 6 hours and advised to take analgesic as needed Aceclofenac, HifinacSR (200 mg); Intas Pharmaceuticals, India. to avoid pain. Patients will also be advised to stop smoking and chewing tobacco products.

Day Two to Three: Routine complete blood investigations including a liver function test (LFT) will be performed at 1 to 2 days following ingestion of ALA. If abnormalities are noted, follow-up blood work will be conducted that includes a renal function test (blood urea, serum creatinine, uric acid) and blood electrolytes measurement.

Day Seven to Ten: At a follow-up examination, 7 days after treatment, an ultrasound of the oral cavity will be conducted to assess treatment response by lesion area (cm2) and depth (mm). As part of this study, ALA will also be re-administered (unless a particular patient had an adverse reaction to ALA in the initial treatment) so that follow-up fluorescence imaging can also be conducted. Again, at this stage, fluorescence imaging is included for validation of the procedure itself, not to decide the next steps in treatment for this patient cohort. However, the follow-up ultrasound will be a decision point to determine whether a given patient needs to undergo surgical excision of residual tumor (possibly with additional radio- and/or chemotherapy as determined by the clinician team), or if no residual disease is present, a biopsy will be conducted at the original disease site for histological confirmation of treatment response, and/or disease progression (development of invasive disease). If the radiologist reports residual tumor after the ultrasound procedure, an ENT surgeon will perform a biopsy and the tissue will be preserved in formalin and sent for histopathology assessment. The depth of necrosis evaluated from the histopathology will serve as endpoint for evaluating the technology. This histopathology data will also be used for validation of imaging to establish fluorescence contrast agreement with histologically confirmed malignant tissue.

Follow-up Model: Patients who have a good response to PDT will not need to undergo surgery, which would compromise the excellent healing of the mucosa that has been reported with this modality. At the same time, patients whose disease has partial or no response to PDT will still receive the same standard of care (surgical excision, chemo/radiation) they would have if they had not enrolled in the study. It is also possible that the PDT treatment, even if the response was not complete, could reduce the scope of excision required in these subjects. Therefore at the end of the study, we will have established the utility of this technology without interrupting the flow of treatment/management of the patients whose disease has partial or no response to PDT. Regardless of the flow of this study, additional follow-up on all patients will be carried out at 1 month,3 months, 6 months, 9 months,12 months, and 2 years after treatment. All patient data obtained will be appropriately de-identified as per local institutional guidelines before off-site analysis, which will continue throughout the study.

The clinical validation study will also serve as an opportunity to gather patient data that will be invaluable in two capacities 1) to obtain important information immediately relevant to individual patient care and 2) with a mind toward sustainability, investigators will seek to understand cultural barriers to acceptance or compliance with the proposed PDT treatment that will be accounted for in outreach and training plans. The present validation study is not powered to make a comparison between different interventions, but rather to provide a validation that the safety and efficacy of the low-cost approach is equivalent to previous reports of PDT treatment for oral cancer in traditional medical settings at JNMC.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 21 years, males or females
2. Subject has read and signed a written informed consent form
3. Subject is willing to have ALA administered and wait for 2-3 hours
4. Subject is willing to receive red light irradiation in the mouth via the fiber probe/applicator and is willing to have the fiber probe/applicator in the mouth for a maximum time of 1 hour
5. Subject is willing to allow investigators to take measurements using smart phone imaging before, during and after light treatment
6. After the procedure, the subject is willing to avoid spicy, hot, or oily foods for at least 6 hours
7. Subject willing to wear full sleeve shirt and full-length garments for couple of hours

Exclusion Criteria:

1. Pregnancy or nursing (ALA is a drug that belongs to FDA pregnancy category C).
2. History of photosensitivity diseases (e.g., lupus erythematosus, porphyrias).
3. Therapy with any photosensitizing medication, e.g., thiazides (for the treatment of high blood pressure), fluoroquinolones, griseofulvin, or sulfonamides (for the treatment of infections), sulfonylureas (for the treatment of diabetes), phenothiazines (for the treatment of emotional problems), and other medications reported to cause photosensitivity within the last 6 months.
4. Subject is unable or unwilling to comply with the study requirements.
5. Subject has any conditions or scars within the location of the test sites that may interfere with the treatment or evaluation.
6. Allergy to porphyrins or ALA.
7. Subject has received laser treatment within 6 months in the area of the treatment.
8. Subject is participating in other potentially confounding research, e.g., currently enrolled in a clinical study of any other unapproved investigational drug or device.
9. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study.
10. Subject has inadequate organ function.
11. Subject has co-morbid systemic illnesses or severe concurrent disease.
12. Subject is being treated for vascular disease.
13. Subject is an employee of the participating sites directly supervised by the investigator.
14. Subject with invasive deep carcinoma evaluated by biopsy.
15. Subject is currently being treated for other cancers with medical or radiation therapy.
16. Subject has AIDS or other infectious diseases, including tuberculosis, hepatitis or herpetic lesions (oral herpes).
17. Subject has oral submucous fibrosis (OSF) resulting in a patient inability to comfortably hold the light applicator in mouth.
18. Subject has Human papillomavirus (HPV) positive tumor.
19. Subject has the tumor at Oropharynx area.
20. We will excludes the patients of the all other oral lesions at sites except: the gingivobuccal sulcus, cheek, floor of the mouth and tongue.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tayyaba Hasan, PhD, Principal Investigator — Massachusetts General Hospital, Boston
Locations (1):
- J.N. Medical College, Aligarh Muslim University, Aligarh, Uttar Pradesh, India

REFERENCES:
- [Derived] Siddiqui SA, Siddiqui S, Hussain MAB, Khan S, Liu H, Akhtar K, Hasan SA, Ahmed I, Mallidi S, Khan AP, Cuckov F, Hopper C, Bown S, Celli JP, Hasan T. Clinical evaluation of a mobile, low-cost system for fluorescence guided photodynamic therapy of early oral cancer in India. Photodiagnosis Photodyn Ther. 2022 Jun;38:102843. doi: 10.1016/j.pdpdt.2022.102843. Epub 2022 Mar 31. PMID 35367616

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were evaluated at the Jawaharlal Nehru Medical College Hospital (JNMC), Aligarh, India, and at ambient remote region outpatient department (OPD) camps. Patients were enrolled if interested following exclusion and inclusion criteria.
Pre-assignment Details: Patients with oral lesions were screened by Ultrasound and histopathological cancer confirmation. Once a patient's oral lesion size and depth were confirmed, he/she was assigned for an oral PDT study.
Groups:
- Aminolevulinic Acid (ALA) Photodynamic Therapy (PDT): Aminolevulinic Acid (ALA) administration, Photodynamic Therapy (PDT) treatment using LED (Light-emitting diode) light source and follow-up.
Period: Overall Study
Arm/Group | Aminolevulinic Acid (ALA) Photodynamic Therapy (PDT)
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aminolevulinic Acid (ALA) Photodynamic Therapy (PDT)
Number analyzed (Participants) | 30
Age, Customized [Number; unit: years]
  21-30 years | 2
  31-40 years | 13
  41-50 years | 7
  51-60 years | 6
  61-70 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  South-Asian | 30
Region of Enrollment [Number; unit: participants]
  India | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Residual Tumor Following Photodynamic Therapy (PDT)
Description: Histologically confirmed the absence of residual disease at follow-up lesion site biopsy (7 days) and from additional clinical examinations during follow-up visits. The follow-up visits happened approximately once every 3 months after treatment until Institutional Review Board (IRB) approval (October 12, 2020).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aminolevulinic Acid (ALA) Photodynamic Therapy (PDT)
Number analyzed (Participants) | 30
Participants | 22

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Aminolevulinic Acid (ALA) Photodynamic Therapy (PDT)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 10/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aminolevulinic Acid (ALA) Photodynamic Therapy (PDT) (N=30)
Discomfort during light treatment (General disorders) | 2
Difficulty in holding PDT applicator in patient mouth (General disorders) | 2
Hypotensive after light treatment (PDT treatment day) (General disorders) | 1
Nausea and vomiting after light treatment (General disorders) | 4
Mild headache after light treatment (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT03638622/Prot_SAP_001.pdf